CLINICAL TRIAL: NCT02761850
Title: Developmental Profile of Ocular Refraction in Patients With Congenital Cataract: A Prospective Cohort Study
Brief Title: Developmental Profile of Ocular Refraction in Patients With Congenital Cataract
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-2
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of prospective cohort study is to describe the developmental profile of refraction change in a large cohort of Chinese CC patients. The decisive factors to the range of myopic shift in unilateral CC appeared to be different from that in bilateral CC, indicating dramatic differences in the etiopathogenesis and refractive prognosis between bilateral and unilateral CC.

DETAILED DESCRIPTION:
The refractive status is crucial to visual function and may change throughout life. For patients with congenital cataract (CC), the developmental profile of refraction is complicated due to the potential influences of diverse clinical manifestations and various treatments, and has not yet been fully characterized.

The investigator described the developmental profile of refraction change in a large cohort of Chinese CC patients. The decisive factors to the range of myopic shift in unilateral CC appeared to be different from that in bilateral CC, indicating dramatic differences in the etiopathogenesis and refractive prognosis between bilateral and unilateral CC. The refraction data from CC patients provided in the study are of clinical significance to the guidelines for CC treatment, especially for IOL calculation concerning the laterality of CC.

ELIGIBILITY:
Inclusion Criteria:

* Children with uncomplicated surgeries
* Children with unilateral/bilateral cataract

Exclusion Criteria:

* Corneal diseases
* Lens luxation
* Glaucoma
* Retinal diseases
* Nystagmus and nanophthalmos

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CC were enrolled from the Childhood Cataract Program of the Chinese Ministry of Health (CCPMOH). The study involved 1,164 participants (6,585 persontimes) enrolled from Jan 2010 to Oct 2015. Cataract removal and/or intraocular lens (IOL) implantation were conducted by two experienced cataract surgeons for participants.
Sampling Method: Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The refraction status (presented as spherical equivalent, SE) | Baseline
  Refractions were conducted with objective retinoscopy and cycloplegia, and performed by experienced optometrists.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lin H, Long E, Chen W, Liu Y. Documenting rare disease data in China. Science. 2015 Sep 4;349(6252):1064. doi: 10.1126/science.349.6252.1064-b. No abstract available. PMID 26339020
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/